CLINICAL TRIAL: NCT04695028
Title: Data Collection for the Constitution of an Observatory for Patients Suffering From Microcrystalline Rheumatism With Morphological Phenotyping
Brief Title: CRYSTALILLE Cohort: Getting the Whole Picture of Crystal-related Arthropathies
Acronym: CRYSTALILLE
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: RC-P00101
Record Dates: First submitted 2020-12-16; First posted 2021-01-05 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Gout; Chondrocalcinosis; Hydroxyapatite
Keywords: Gout; Chondrocalcinosis; Hydroxyapatite
MeSH Terms: conditions — Gout; Chondrocalcinosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons with crystal related arthropathies
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — The following data will be collected by the physician: sociodemographic profile, clinical manifestations, comorbidities, laboratory tests,etc.
  Diagnostic performance of different imagery techniques, performance of crystal deposit quantification in ultrasound and Dual-energy computed tomography (DECT), link between co-morbidities and volume of baseline crystal deposits then during monitoring, link between co-morbidities (including cardiovascular events and new diagnoses of co-morbidity) and vascular baseline crystal deposits and during follow-up, link between microcrystalline rheumatism activity and the quantity of crystal deposits in baseline imaging and during follow-up, link between co-morbidities and the evolution of microcrystalline baseline rheumatism and then during follow-up, link between co-morbidities and the evolution of crystal deposition volumes, the concordance of the evaluation of uratic stocks and their evolution between the imagery means.

SUMMARY:
The objective of this research is to collect data to create an observatory of microcrystalline rheumatism (gout and calcium-crystal rheumatism) in patients treated at the Groupement des Hôpitaux de l'Institut Catholique de Lille, in order to better understand the disease and improve patient care, in particular with the help of medical imaging.

DETAILED DESCRIPTION:
All patients already included in another observational study set up in 2016 and meeting the eligibility criteria may be included in this study. An information letter will be sent to them by mail. If they wish to oppose to the use of their data, they can then return the objection form.

This sample will be supplemented by new patients who are recruited during a classic rheumatology consultation. The investigator will propose the study to all patients meeting the inclusion and non-inclusion criteria.

They will be informed of the objectives of the study and their rights. For patients who agree to participate in the study, sociodemographic and clinical characteristics will be collected.

Depending on the usual care, they will benefit from an ultrasound and/or a dual energy scanner (M0). Imaging data will be collected. Routine clinical follow-up is then carried out in consultation, with collection of clinical and biological evolution data, and morphological data if necessary if imaging is rechecked, until the patient is lost to follow-up or the follow-up is interrupted at the GHICL for any reason.

Available quarterly or semi-annual data will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gout according to American College of Rheumatology /European League Against Rheumatism (ACR/EULAR) 2015 criteria OR diagnosis of calcium pyrophosphate dihydrate crystal deposition disease (CPPD) based on EULAR 2011 recommendations OR diagnosis of hydroxyapatite crystal rheumatism (HCR) according to a typical clinical sequence and demonstration of compatible calcium deposits on imaging
* patient who will benefit or has benefited from an ultrasound and/or DECT evaluation of microcrystalline deposits
* clinical suspicion of microcrystalline rheumatism requiring further imaging to confirm the diagnosis

Exclusion Criteria:

* Refusal or contra-indication to perform ultrasound or dual energy scanning.
* Patient's opposition to the use of his or her health data for research purposes
* Patient under guardianship or curatorship
* Pregnant woman
* Person not affiliated to a social security scheme or entitled to a social security benefit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gout Chondrocalcinosis Hydroxyapatite
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of microcrystalline rheumatism | day 0
Weight | day 0
  measured in Kg
Height | day 0
  measured in cm
Index body mass | day 0
Comorbidities | day 0
Number of rheumatic flares | day 0
Intensity of rheumatic flares | day 0
Identification of subcutaneous tophi | day 0
Uricemia | day 0
Renal function panel | day 0
  Panel includes albumin, calcium, carbon dioxide, creatinine, chloride, glucose, phosphorous, potassium, sodium, and BUN and a calculated anion gap value
Lipid profile | day 0

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Pascart, MD, Principal Investigator — GHICL
Locations (1):
- GHICL- Hôpital Saint Philibert, Lomme, France

IPD SHARING:
Plan to Share IPD: Yes